CLINICAL TRIAL: NCT04693936
Title: Study of Metabolic Pathways for the Identification of Biomarkers in Hashimoto's Thyroiditis and Psoriasis
Brief Title: Metabolic Biomarkers in Hashimoto's Thyroiditis and Psoriasis
Acronym: METHAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Evangelia Sarandi, Biologist, MSc, PhD student, University of Crete
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 147/26.06.2020
Record Dates: First submitted 2020-12-23; First posted 2021-01-05 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Hashimoto Disease; Psoriasis
Keywords: metabolomics; biomarkers; metabolic pathways
MeSH Terms: conditions — Hashimoto Disease; Psoriasis

STUDY DESIGN:
Intervention Model Description: Patients with Hashimoto's disease and patients with psoriasis and healthy individuals will be randomly assigned to intervention group and to control group. The intervention will be a nutraceuticals supplements combination in the context of Mediterranean diet. The duration of the intervention will last 6 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutraceuticals (Active Comparator): Participants will receive a combination of nutraceuticals and will be instructed to follow a Mediterranean diet
  Interventions: Combination Product: Nutraceutical Combination Plan
- Control (No Intervention): Participants will follow usual diet

INTERVENTIONS:
Combination Product: Nutraceutical Combination Plan — Multivitamin (My Total Health) 1 tablet per day Vitamin C (My Immuno) 1 scoop per day Calcium-Magnesium combination (My Calmag) 1 scoop per day Omega 3-6-9 My Omega Krill. 1 capsule per day Glutamine (L-Glutamin &Chios Mastiha) 1 tablet per day Probiotics 40 billion 1 capsule per day
  Nutraceuticals will be received daily along with the patient's customary psoriasis/Hashimoto's disease treatment.
  Arms: Nutraceuticals

SUMMARY:
Hashimoto's disease (HT) and psoriasis (PsO) have a significant impact on patient's quality of everyday life, and early diagnosis is critical for the symptoms management and prognosis. There is evidence that HT and PsO share common metabolic pathways that relate to their pathogenesis, and are affected by dietary and lifestyle factors. Previous studies have identified potential metabolic biomarkers, although the small number of studies hamper their validation. Of note, most studies are not longitudinal thus do not capture the metabolic fluctuations in response to disease progression or dietary changes. Thus, the purpose of this study is to identify metabolic biomarkers of HT and PsO and study the role of epigenetic factors (diet and lifestyle) on the involved metabolic pathways . In addition, a comparative analysis of the disease-related quality of life (QoL) will be performed in relation to dietary changes to unravel possible links between the QoL and the associated metabolic pathways in HT and PsO.

DETAILED DESCRIPTION:
Patients with Hashimoto's thyroiditis (HT), patients with psoriasis (PsO), and healthy individuals aged 18-60 will be recruited and assessed according to inclusion/exclusion criteria. Eligible participants will be randomized to two groups. The intervention group will receive a combinational nutraceuticals plan for 6 months as part of a Mediterranean diet and the control group will follow usual diet. Data will be collected at baseline and at the end of the study including levels of organic and fatty acids, lifestyle and anthropometric measurements, adherence to Mediterranean diet through the Mediterranean Diet Score (MDS) and disease-specific quality of life through the Thyroid Patient Report Outcome (THYPRO) and the Dermatology Life Quality Index (DLQI) questionnaires for the HT and the PsO group respectively.

ELIGIBILITY:
Hashimoto's Thyroiditis:

* Clinical findings
* Presence of thyroid autoantibodies (anti-TPO) in laboratory tests
* Gray-scale Ultrasound findings.

Psoriasis:

* Presence of psoriatic lesions
* Psoriasis Area and Severity Index score (PASI).

Healthy group:

Non-obese (BMI<30)

* non-athletes
* non-pregnant or lactating women
* not been diagnosed with a chronic or acute disease
* not receiving antidepressants, drugs and supplements
* normal Thyroid Stimulating Hormone (TSH) levels or high TSH and absence of other clinical findings of thyroid malfunction.

Exclusion Criteria:

* malignant or congenital goiter
* thyroidectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Differential levels of urinary organic acids in patients with Hashimoto's thyroiditis and psoriasis compared to healthy individuals as assessed by GC-MS | Baseline
  Levels of organic acids will be quantified in the urine of patients with Hashimoto's diseases and psoriasis and the healthy group at baseline. Concentrations will be calculated in relation to creatinine (mmol/mol Crea) using Gas Chromatography-Mass Spectrometry (GC-MS).
  Comparisons will be made at organic acids concentrations between the HT, the PSO and the healthy group to determine disease-related differences
Differential levels of peripheral blood fatty acids in patients with Hashimoto's thyroiditis and psoriasis compared to healthy individuals as assessed by GC-MS | Baseline
  Levels of total fatty acids will be quantified (μmol/l) in the peripheral blood of patients with Hashimoto's diseases and psoriasis and the healthy group at baseline using Gas Chromatography-Mass Spectrometry (GC-MS)
  Comparisons will be made at fatty acids concentrations between the HT, the PSO and the healthy group to determine disease-related differences
Change from baseline urinary organic acids levels after 6-month intervention with nutraceuticals as assessed by GC-MS | 6 months
  Levels of organic acids will be quantified in the urine of patients with Hashimoto's diseases and psoriasis and the healthy group after 6 months of intervention. Concentrations will be calculated in relation to creatinine (mmol/mol Crea).
  Comparisons will be made at organic acids concentrations between baseline levels and post 6 months treatment in the HT, the PSO and the healthy group to determine intervention-related differences
Change from baseline peripheral blood fatty acids levels after the 6-month intervention with nutraceuticals as assessed by GC-MS | 6 months
  Levels of total fatty acids will be quantified (μmol/l) in the peripheral blood of patients with Hashimoto's diseases and psoriasis and the healthy group after 6 months of intervention.
  Comparisons will be made at fatty acids concentrations between baseline levels and post 6 months of treatment in the HT, the PSO and the healthy group to determine intervention-related differences
Change from baseline thyroid disease-related quality of life at 6-months of intervention with nutraceuticals as assessed by the THYPRO questionnaire | 6 months
  The Thyroid Patient Response Outcome (THYPRO) questionnaire will be completed by the HT group at baseline and 6 months post intervention (both arms).
  THYPRO score (0-100) after the intervention will be compared with baseline.
Change from baseline psoriasis-related quality of life at 6-months of intervention with nutraceuticals as assessed by the DLQI questionnaire | 6 months
  The Dermatology Life Quality Index (DLQI) will be completed by the HT group and the PSO group (both arms) at baseline and 6 months post intervention.
  DLQI score (0-30) after the intervention will be compared with baseline.
Change from baseline Mediterranean diet adherence at 6 months of intervention with nutraceuticals as assessed by the MDS questionnaire | 6 months
  The Mediterranean Diet Score (MDS) questionnaire will be collected for all participants (both arms) at baseline and 6 months post the intervention.
  MDS (0-17) after the intervention will be compared with baseline.

SECONDARY OUTCOMES:
Change from baseline Body Mass Index at 6 months of intervention with nutraceuticals | 6 months
  BMI will be estimated at baseline and 6 months post the intervention for the three groups (both arms).
  For the estimation of BMI (kg/m^2) weight and height will be combined
Change from baseline waist circumference at 6 months of intervention with nutraceuticals | 6 months
  Waist circumference (cm) will be measured at baseline and 6 months post the intervention for the three groups (both arms).
Change from baseline alcohol consumption at 6 months of intervention with nutraceuticals | 6 months
  Alcohol consumption (number of glasses per week) will be assessed at baseline and 6 months post the intervention for all participants (both arms).
Change from baseline physical activity at 6 months of intervention with nutraceuticals | 6 months
  Physical activity frequency (times per week) will be assessed at baseline and 6 months post the intervention for all participants (both arms).
Change from baseline smoking at 6 months of intervention with nutraceuticals | 6 months
  Smoking (cigars per day) will be assessed at baseline and 6 months post the intervention for all participants(both arms).

CONTACTS AND LOCATIONS:
Overall Officials: Aristidis Tsatsakis, PhD, Prof, Study Chair — University of Crete; Sabine Kruger-Krasagakis, MD,Ass Prof, Principal Investigator — University of Crete; Gottfried Rudofsky, MD, Prof., Principal Investigator — Heidelberg University
Locations (1):
- Metabolomic Medicine, Private Health Clinics, Athens, Greece

IPD SHARING:
Plan to Share IPD: No